CLINICAL TRIAL: NCT02009839
Title: Effectiveness of a Web-Based CBT Protocol for Treatment of Selective Mutism in Singapore
Brief Title: Web-Based CBT Protocol for Treatment of Selective Mutism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Healthcare Group, Singapore (Other Government)
Responsible Party: Principal Investigator, A/Prof Daniel Fung Shuen Sheng, Dr, National Healthcare Group, Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NHG-SIG/05016
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Selective Mutism
Keywords: anxiety; frequency of speech; selective mutism
MeSH Terms: conditions — Mutism; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meeky Mouse program (Experimental): 14-week "Meeky Mouse" program consists of 8 training sessions (psychoeducation and anxiety management) followed by 6 practice sessions (exposure using social skills training)
  Interventions: Behavioral: Meeky Mouse program
- Computer Games (Placebo Comparator): 14 weeks of interactive session with the therapist while playing computer games
  Interventions: Other: Computer Games

INTERVENTIONS:
Behavioral: Meeky Mouse program
  Arms: Meeky Mouse program
Other: Computer Games
  Arms: Computer Games

SUMMARY:
The main aim of this study is to examine the effectiveness of a web-based CBT protocol (entitled Meeky Mouse) in the treatment of children with Selective Mutism in Singapore. The researchers hypothesized that the Meeky Mouse program would be associated with higher frequency of speaking behaviors, lower levels of anxiety, greater improvements in clinician-rated severity of mental illness, and higher clinician-rated improvement scores at post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* 6-12 years old
* primary clinical diagnosis of Selective Mutism
* confirmed diagnosis of Selective Mutism by structured clinical parent interview
* fluent in English

Exclusion Criteria:

* below average intellectual functioning
* the presence of autism and schizophrenia

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2005-07; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Selective Mutism Questionnaire | Changes from pre-treatment (Week 0) to post-treatment (Week 14) on SMQ scores

SECONDARY OUTCOMES:
Asian Children's Anxiety Scale-Caretaker Version (ACAS) | Changes from pre-treatment (Week 0) to post-treatment (Week 14) on ACAS total scores
Asian Children's Anxiety Scale-Child (ACAS-C) | Changes from pre-treatment (Week 0) to post-treatment (Week 14) on ACAS-C total scores
Clinical Global Impression (CGI) | Changes from pre-treatment (Week 0) to post-treatment (Week 14) on CGI-Severity and CGI-Improvement Ratings

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fung, MBBS, MMed, Principal Investigator — Institute of Mental Health, Singapore
Locations (1):
- Child Guidance Clinic, Singapore, Singapore